CLINICAL TRIAL: NCT05445583
Title: Asthma and Technology in Emerging African American Adults (The ATHENA Project).
Brief Title: Asthma and Technology in Emerging African American Adults
Acronym: ATHENA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Alan Baptist, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01NR019566 (NIH); 1R01NR019566-01A1 (NIH)
Record Dates: First submitted 2022-04-14; First posted 2022-07-06 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Asthma
Keywords: African American; Young Adult; eHealth; Mobile Health
MeSH Terms: conditions — Asthma | interventions — Spermine Synthase

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Motivational Enhancement System (MES) and Physical Activity Tracking (PAT) (Experimental): MES is a web-based, mobile asthma management intervention delivered to participants' personal mobile devices. There are 4 sessions, completed over 10 weeks, with each session taking approximately 15-20 minutes. During Session 1, participants will identify asthma-related problems they may encounter and will receive asthma information and motivation. Between Session 1 and Session 2, participants will be asked to complete an electronic daily diary for 7 days. Session 2 allows participants to select up to 2 goals to address. Session 3 occurs over the course of 4 weeks and provides tailored messages based on problem and goal selection. The final session (Session 4), asks participants for feedback on how well they feel they accomplished their goal. Additionally, participants will be asked to track their daily and weekly step totals as well their total minutes of moderate to vigorous physical activity using a wearable activity tracker provided by the study.
  Interventions: Behavioral: Motivational Enhancement System (MES); Behavioral: Physical Activity Tracking (PAT)
- Supportive Accountability (SA) and PAT (Experimental): SA is an asthma management intervention delivered by asthma nurses trained in targeted MI skills (e.g., open-ended questions around change talk, affirmations) via participants' personal mobile devices (e.g., Skype, FaceTime, voice calls, and SMS). Sessions with the nurse will be approximately 15-20 minutes in length and will focus on ways to improve asthma care. There are 4 sessions with the nurse, over the course of 10 weeks. Additionally, participants will be asked to track their daily and weekly step totals as well their total minutes of moderate to vigorous physical activity using a wearable activity tracker provided by the study.
  Interventions: Behavioral: Supportive Accountability (SA); Behavioral: Physical Activity Tracking (PAT)
- Text Messaging (SMS) and PAT (Experimental): SMS will target asthma knowledge. One-way SMS messages will be sent to participants' personal mobile devices with facts about asthma management, links to educational web content, and videos providing information about living with asthma. Text messages will be sent twice a week for the first 5 weeks and once a week for the last 5 weeks. Additionally, participants will be asked to track their daily and weekly step totals as well their total minutes of moderate to vigorous physical activity using a wearable activity tracker provided by the study.
  Interventions: Behavioral: Motivational Enhancement System (MES); Behavioral: Physical Activity Tracking (PAT)
- MES_SMS_PAT (Experimental): Participants will receive a combination of the MES and SMS interventions. Additionally, participants will be asked to track their daily and weekly step totals as well their total minutes of moderate to vigorous physical activity using a wearable activity tracker provided by the study.
  Interventions: Behavioral: Motivational Enhancement System (MES); Behavioral: Text Messaging (SMS); Behavioral: Physical Activity Tracking (PAT)
- SA_SMS_PAT (Experimental): Participants will receive a combination of the SA and SMS interventions. Additionally, participants will be asked to track their daily and weekly step totals as well their total minutes of moderate to vigorous physical activity using a wearable activity tracker provided by the study.
  Interventions: Behavioral: Motivational Enhancement System (MES); Behavioral: Text Messaging (SMS); Behavioral: Physical Activity Tracking (PAT)
- Usual Care_PAT (No Intervention): Participants will continue to receive standard clinical asthma care. Additionally, participants will be asked to track their daily and weekly step totals as well their total minutes of moderate to vigorous physical activity using a wearable activity tracker provided by the study.

INTERVENTIONS:
Behavioral: Motivational Enhancement System (MES) — MES is an eHealth application and focuses on asthma management behaviors with feedback on asthma symptoms, physical activity, adherence, and tailored education. The program is interactive and tailored to each participant by (1) allowing participants to choose barriers/goals related to their asthma care and (2) by sending personalized feedback based on participant daily diary responses. MES consists of 4 sessions delivered over the course of 10 weeks within 10 smaller 5-10 minute blocks.
  Arms: MES_SMS_PAT; Motivational Enhancement System (MES) and Physical Activity Tracking (PAT); SA_SMS_PAT; Text Messaging (SMS) and PAT
Behavioral: Supportive Accountability (SA) — Supportive accountability (SA) is an asthma management intervention delivered by asthma nurses trained in motivational interviewing skills (e.g., open-ended questions around change talk, affirmations) via participants' personal mobile devices (e.g., Skype, FaceTime, voice calls, and SMS). The theory underlying SA is that education and behavior change are most impactful when delivered by a knowledgeable yet supportive authority figure (i.e. nurse).
  Arms: Supportive Accountability (SA) and PAT
Behavioral: Text Messaging (SMS) — SMS will target asthma knowledge. SMS messages will be sent via CIAS 3.0 to participants' personal mobile devices with facts about asthma management, links to educational web content, and videos providing information about living with asthma. Information covered includes 'What is asthma,' 'What is an asthma attack,' 'What causes an asthma attack,' 'How is asthma treated,' 'Asthma and weather,' 'Using an inhaler,' 'Using a spacer,' and 'Asthma Action Plans.'
  Arms: MES_SMS_PAT; SA_SMS_PAT
Behavioral: Physical Activity Tracking (PAT) — All participants will be provided a wearable physical activity tracking device, which will allow them to accurately track exercise and total steps each day. Through PAT, users will be able to set daily goals and attain motivation to continue asthma management. For individuals randomized to groups that also include MES or SA, those programs will incorporate PAT data that is remotely transmitted, to facilitate asthma management motivation.
  Arms: MES_SMS_PAT; Motivational Enhancement System (MES) and Physical Activity Tracking (PAT); SA_SMS_PAT; Supportive Accountability (SA) and PAT; Text Messaging (SMS) and PAT

SUMMARY:
The purpose of the ATHENA Project is to test a mobile health intervention to help African American young adults better manage their asthma. The program has four components: 1) a web-based, mobile asthma program delivered to participants' mobile device, 2) meetings with an asthma nurse via video conference, 3) text messaging, and 4) physical activity tracking. Participants will be randomly assigned to one or more of these components to better meet the needs of young adults with asthma.

DETAILED DESCRIPTION:
Asthma causes substantial morbidity and mortality in the United States, particularly among African American emerging adults (AAEA; ages 18-30), but very few asthma programs have targeted this population. Interventions that provide education and address underlying motivation for managing asthma may be most effective. However, face-to-face interventions are often difficult to implement, especially among emerging adults. Mobile asthma management interventions may help improve asthma control and allow people to live healthier lives. During this project, the research team will use an innovative strategy to develop a mobile asthma management intervention using the most effective combination of a smart phone app delivering personalized asthma information (MES), nurse-delivered asthma education (SA), text messaging (SMS), and physical activity tracking (PAT).

The purpose of this proposal is to develop an effective mHealth intervention to improve asthma management and asthma control in AAEA. Investigators will assess the ability of multiple technologic components to assist and improve traditional asthma education. Upon completion of the study, investigators will have an empirically-supported mobile asthma management intervention to improve asthma control for AAEA.

It is hypothesized that post-intervention, participants with uncontrolled asthma will show clinically-significant improvement in asthma control and improvements in asthma management behaviors, quality of life, symptoms, adherence, and exacerbations will also be observed.

ELIGIBILITY:
Inclusion Criteria:

* African American, 18-30 years of age, uncontrolled asthma (defined by a score of less than 19 on the ACT), own or have access to a cell phone for the duration of the study, have a primary care physician (PCP)

Exclusion Criteria:

* Significant cardiopulmonary disease (including chronic obstructive pulmonary disease), a greater than 20 pack per year smoking history, developmental delay or mental illness such that participation in the program would not be possible, pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Test (ACT) | Change from baseline at 3, 6, and 12 months
  Frequency of asthma symptoms based on self-report

SECONDARY OUTCOMES:
Asthma Quality of Life Questionnaire (AQLQ) | Change from baseline at 3, 6, and 12 months
  Measures functional impairments that are most troublesome to adults with asthma
Asthma exacerbations | Change from baseline at 3, 6, and 12 months
  Reduction in number of asthma exacerbations
Medication Adherence Report Scale for Asthma (MARS-A) | Change from baseline at 3, 6, and 12 months
  Self reported adherence to asthma controller medication
International Physical Activity Questionnaire (IPAQ) | Change from baseline at 3, 6, and 12 months
  Assess kinds of physical activities and time spent being physically active

CONTACTS AND LOCATIONS:
Overall Officials: Alan Baptist, MD., Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - Florida State University, Tallahassee, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No